CLINICAL TRIAL: NCT03406689
Title: Comparison of the Efficacy of Nepafenac 0.1% and Nepafenac 0.3 % on Pain Associated With Intravitreal Injections, a Triple Arm Study
Brief Title: Comparison of the Efficacy of Nepafenac 0.1% and Nepafenac 0.3 % on Pain Associated With Intravitreal Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Constantinos D. Georgakopoulos, MD, PhD, Associate Professor in Ophthalmology, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 72/15.04.2016
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Pain
Keywords: Pain; Intravitreal Injection; Anti-VEGF; Nepafenac eye drops; Short Form McGill Pain Questionnaire
MeSH Terms: conditions — Pain | interventions — nepafenac; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nepafenac 0.1% Oph Susp (Active Comparator): One drop of Nepafenac 0.1% will be administered 45' prior to the injection
  Interventions: Drug: Nepafenac 0.1% Oph Susp
- Nepafenac 0.3% Oph Susp (Active Comparator): One drop of Nepafenac 0.3% will be administered 45' prior to the injection
  Interventions: Drug: Nepafenac 0.3% Oph Susp
- Artificial tears (Placebo Comparator): One drop of Artificial Tears will be administered 45' prior to the injection
  Interventions: Drug: Artificial tear

INTERVENTIONS:
Drug: Nepafenac 0.1% Oph Susp — One drop of Nepafenac 0.1% will be instilled 45' prior to the IVI.
  Other Names: NEVANAC EY.DRO.SUS 1MG/ML
  Arms: Nepafenac 0.1% Oph Susp
Drug: Nepafenac 0.3% Oph Susp — One drop of Nepafenac 0.3% will be instilled 45' prior to the IVI.
  Other Names: NEVANAC EY.DRO.SUS 3MG/ML
  Arms: Nepafenac 0.3% Oph Susp
Drug: Artificial tear — One drop Artificial Tears will be instilled 45' prior to the IVI.
  Other Names: TEARS NATURALE EY.DRO.SOL 0,1%+0,3%
  Arms: Artificial tears

SUMMARY:
The analgestic efffect of Nepafenac 0.1% Eye Drops and Nepafenac 0.3% Eye Drops on pain related to intravitreal injections will be evalutated.

Pain perception will be assessed by the Short Form of the McGill Pain Questionnaire.

DETAILED DESCRIPTION:
Intravitreal injection (IVI) is a preferred route of administration of drugs in the posterior segment of the eye. Intravitreal injection of anti-VEGFs constitutes the mainstay for the treatment of various retinal diseases such as AMD, RVO, DME etc. The procedure of the IVI is, however, associated with a level of discomfort for the patient.

Nonsteroidal anti-inflammatory drugs (NSAIDs) inhibit the activity of cyclooxygenase-1 and cyclooxygenase-2, and thereby, the synthesis of prostaglandins and thromboxanes. Cyclooxygenase-2 inhibition leads to the anti-inflammatory, analgesic and antipyretic effects of NSAIDs. Ophthalmic NSAIDs constitute an established and effective treatment option for the management of inflammation and pain associated with cataract surgery and of pain associated with corneal refractive surgery, for inhibition of intraoperative miosis and for the treatment of seasonal allergic conjunctivitis.

The primary goal of this study is to assess the analgesic effect of Nepafenac 0.1% and Nepafenac 0.3% Eye Drops on pain related to intravitreal injections immediately after and up to six hours postIVI.

A number of patients scheduled to undergo IVIs of anti-VEGFs will be randomized and divided in three groups. All patients must have already undergone at least one IVI. In patients receiving IVIs in both eyes only one eye will be included in the study.

The patients of the first group will receive Nepafenac 0.1 % Eye Drops 45 minutes prior to the injection.

The patients of the second group will recieve Nepafenac 0.3 % Eye Drop 45 minutes prior to the injection. The patients of the third group will receive Artificial Tears 45 minutes prior to the injection.

Patients will be required to complete the greek version of the short form McGill Pain Questionnaire (SF-MPQ) comprising of the Visual Analogue Scale, the main component of the SF-MPQ and the Present Pain Intensity Scale immediately after the injection and 6 hours post-IVI.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be patients of the Medical Retina Department of our Clinic, who are scheduled to receive IVIs of ranibizumab (Lucentis; Novartis Pharma S.A.S., Huningue, France) or aflibercept (Eylea; Bayer Healthcare Pharmaceuticals, Berlin, Germany) in one eye and had already undergone at least one IVI of an anti-VEGF agent.

Exclusion Criteria:

* History of previous eye surgery other than cataract extraction surgery, herpetic eye disease, uncontrolled glaucoma, uveitis, active conjunctivitis, keratitis and bullous keratopathy, a previously known allergic response to nepafenac or other NSAIDs and salicylates, any contraindication to NSAIDs administration such as cardiovascular disease, gastrointenstinal disease with risk of GI ulceration,bleeding and perforation, renal and hepatic disease and any systemic or topical use of NSAIDs or any use of sedative medications within 7 days from the visit and during the day of IVI.
* Patients with poor cooperation in understanding and answering the questions of the SF-MPQ, including the visual analogue scale (VAS).
* Unsuccessful blinding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Assessment of topical Nepafenac 0.1% and Nepafenac 0.3% analgesic effect in patients undergoing intravitreal injections of anti-VEGFs | Immediately after the injection
  As measured by the Visual Analogue Scale. The Visual Analogue Scale (abbreviation VAS) is a self report pain score chart designed as a 10 cm horizontal line marked at both ends. Each boundary of the line represents the extremes of painful experience (0=no pain and 10= the worst pain ever experienced).
  The patient is asked to mark on the scale the exact point corresponding to their perception of pain intensity and the score is calculated by measuring from the left hand side to the mark made by the patient, ranging from 0 to 10.
  Higher scores indicate more severe pain.

SECONDARY OUTCOMES:
Assessment of topical Nepafenac 0.1% and Nepafenac 0.3% analgesic effect in patients undergoing intravitreal injections of anti-VEGFs | Six hours after injection
  As measured by the Visual Analogue Scale. The Visual Analogue Scale (abbreviation VAS) is a self report pain score chart designed as a 10 cm horizontal line marked at both ends. Each boundary of the line represents the extremes of painful experience (0=no pain and 10= the worst pain ever experienced).
  The patient is asked to mark on the scale the exact point corresponding to their perception of pain intensity and the score is calculated by measuring from the left hand side to the mark made by the patient,ranging from 0 to 10.
  Higher scores indicate more severe pain.
Assessment of topical Nepafenac 0.1% and Nepafenac 0.3% analgesic effect in patients undergoing intravitreal injections of anti-VEGFs | Immediately after the injection
  As measured by the Main Component of the Short Form of the McGill Pain Questionnaire.
  The main component of the Short form of the McGill Pain Questionnaire (abbreviation SF-MPQ) comprises of 15 adjectives describing the pain experienced (11 sensory and 4 affective). The patient is asked to grade the intensity of each specific pain quality on an intensity scale from 0 to 3 (0= none, 1=mild, 2=moderate, 3=severe).
  The total score of the main component is derived by adding the rank values given by the patient for each descriptor out of 45. Scores can range from 0 to 45.
  A higher score of the main component of the SF-MPQ reflects more serious pain.
Assessment of topical Nepafenac 0.1% and Nepafenac 0.3% analgesic effect in patients undergoing intravitreal injections of anti-VEGFs | Six hours after injection
  As measured by the Main Component of the Short Form of the McGill Pain Questionnaire.
  The main component of the Short form of the McGill Pain Questionnaire (abbreviation SF-MPQ) comprises of 15 adjectives describing the pain experienced (11 sensory and 4 affective). The patient is asked to grade the intensity of each specific pain quality on an intensity scale from 0 to 3 (0= none, 1=mild, 2=moderate, 3=severe).
  The total score of the main component is derived by adding the rank values given by the patient for each descriptor out of 45. Scores can range from 0 to 45.
  A higher score of the main component of the SF-MPQ reflects more serious pain.
Assessment of topical Nepafenac 0.1% and Nepafenac 0.3% analgesic effect in patients undergoing intravitreal injections of anti-VEGFs | Immediately after the injection
  As measured by the Present Pain Intensity score. The PPI index is a numerical verbal rating scale consisting of 6 adjectives of gradually increasing pain sensation (0, none; 1, mild; 2, discomforting; 3, distressing; 4, horrible; and 5, excruciating).
  The patient is instructed to choose the adjective indicating their pain state. The score for the PPI is derived from the number next to the patients' adjective of choice, ranging from 0 to 5.
  Higher scores indicate more intense pain.
Assessment of topical Nepafenac 0.1% and Nepafenac 0.3% analgesic effect in patients undergoing intravitreal injections of anti-VEGFs | Six hours after injection
  As measured by the Present Pain Intensity score. The Present Pain Intensity (abbreviation PPI) index is a numerical verbal rating scale consisting of 6 adjectives of gradually increasing pain sensation (0, none; 1, mild; 2, discomforting; 3, distressing; 4, horrible; and 5, excruciating).
  The patient is instructed to choose the adjective indicating their pain state. The score for the PPI is derived from the number next to the patients' adjective of choice, ranging from 0 to 5.
  Higher scores indicate more intense pain.

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Georgakopoulos, MD, PhD, Principal Investigator — Associate Professor of Ophthalmology, Medical School, University of Patras, Greece
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: Undecided